CLINICAL TRIAL: NCT03789578
Title: A Trial to Investigate Single Dose Pharmacokinetics of NNC0148-0287sema in a Fixed Ratio Compared With Insulin 287 and Semaglutide Given Separately in Subjects With Type 2 Diabetes
Brief Title: A Research Study to Look at How Insulin 287 and Semaglutide Work in the Body of People With Type 2 Diabetes When Taken Alone or Together
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NN1535-4359; U1111-1204-8233 (Other: World Health Organization (WHO)); 2017-004538-27 (Registry Identifier: European Medicines Agency (EudraCT))
Record Dates: First submitted 2018-12-27; First posted 2018-12-28 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — semaglutide

STUDY DESIGN:
Intervention Model Description: This is a three-period cross-over trial. The treatments to be used are: Treatment A: insulin 287, Treatment B: semaglutide, and Treatment C: NNC0148-0287sema. The subjects will be randomised to one of the six treatment sequences in the trial: 1) ABC, 2) ACB, 3) BAC, 4) BCA, 5) CAB, and 6) CBA. The trial includes a screening visit followed by three 5 -week periods with pharmacokinetic sampling after single dose administration. The dose periods are separated by a 1-4 week washout period (from last pharmacokinetic sampling to next dosing). The follow-up period is 1-4 weeks after last pharmacokinetic sampling in period 3 (i.e. 6 to 9 weeks after last trial product administration). The total trial duration for the individual subjects participating in the trial will be 19 to 32 weeks (including follow-up), depending on individual visit schedules.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Sponsor staff involved in the clinical trial is masked according to company standard procedures.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Semaglutide plus insulin 287 (Experimental): Participants will get a single dose of fixed-ratio combination of insulin 287 and semaglutide (NNC0148-0287sema (treatment C)).
  Interventions: Drug: NNC0148-0287sema
- Semaglutide alone (Experimental): Participants will get a single dose of semaglutide (treatment B) alone.
  Interventions: Drug: Semaglutide
- Insulin 287 alone (Experimental): Participants will get a single dose of insulin 287 (NNC0148-0287 (treatment A)) alone.
  Interventions: Drug: NNC0148-0287

INTERVENTIONS:
Drug: NNC0148-0287sema — Study staff will inject NNC0148-0287sema, 175unit (U)/0.5 mg in the morning after fasting under the skin of participants' thigh using a needle and a pen.
  Arms: Semaglutide plus insulin 287
Drug: Semaglutide — Study staff will inject semaglutide, 0.5 mg alone in the morning after fasting under the skin of participants' thigh using a needle and a pen.
  Other Names: Ozempic®
  Arms: Semaglutide alone
Drug: NNC0148-0287 — Study staff will inject insulin 287 (NNC0148-0287), 175U alone in the morning after fasting under the skin of participants' thigh using a needle and a pen.
  Arms: Insulin 287 alone

SUMMARY:
The study will look at how insulin 287 and semaglutide work in the body, both when given alone or together. This study will look at the way insulin 287 and semaglutide reach and stay in participants' blood after injection when given alone or together. Participants will get 3 study medicines at 3 different time points: 1) a combination of semaglutide plus insulin 287, 2) insulin 287 alone and 3) semaglutide alone. The order in which participants get them is decided by chance. Participants will get all medicines as an injection under the skin in the thigh. The injections will be done by study staff. The time between injections is 6 to 9 weeks. The study will last for about 19 to 32 weeks in total.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged 18-64 years (both inclusive) at the time of signing informed consent
* Diagnosed with type 2 diabetes mellitus more than or equal to 180 days prior to the day of screening
* Body weight between 80.0 to 120.0 kg (both inclusive)
* Glycosylated haemoglobin (HbA1c) 6.0 to 8.5% (both inclusive)
* No current and no regular previous intake of insulin. Previous insulin treatment for short periods of time (a maximum of 14 days) is allowed, as well as insulin use during a previous period of gestational diabetes in the past (as declared by the subject or reported in the medical records)
* Stable daily dose(s) of the following anti-diabetic drug(s)/regimen within the past 90 days prior to the day of screening: a) Any metformin formulation (dose as documented in the subject medical record), b) One other oral antidiabetic drug (dose as documented in the subject medical record) is allowed, but not mandatory: Insulin secretagogue (sulphonylureas), dipeptidyl peptidase 4 (DPP-4) inhibitor and sodium glucose co-transporter 2 (SGLT2) inhibitor

Exclusion Criteria:

* Known or suspected hypersensitivity to trial products or related products
* Female who is pregnant, breast-feeding or intends to become pregnant or is of child-bearing potential and not using adequate contraceptive methods
* Recurrent severe hypoglycaemia (more than 1 severe hypoglycaemic event within the past 180 days) or hypoglycaemic unawareness as judged by the investigator or hospitalisation for diabetic ketoacidosis within the past 180 days prior to the day of screening
* Receipt of any investigational medicinal product within 90 days before screening
* History of severe allergies to drugs or foods or a history of severe anaphylactic reaction

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2019-01-17 (Actual); Primary Completion 2019-10-10 (Actual); Study Completion 2019-10-10 (Actual)

PRIMARY OUTCOMES:
AUCI287, 0-tz, area under the serum insulin 287 concentration-time curve from 0 hours to last quantifiable observation after a single dose | 0-840 hours
  Measured in pmol*h/L for insulin 287 following administration of a fixed ratio of NNC0148-0287sema and insulin 287.
AUCSema,0-tz, area under the plasma semaglutide concentration-time curve from 0 hours to last quantifiable observation after a single dose | 0-840 hours
  Measured in pmol*h/L for semaglutide following administration of a fixed ratio of NNC0148-0287sema and semaglutide.

SECONDARY OUTCOMES:
AUCI287,0-∞ area under the serum insulin 287 concentration-time curve from 0 hours to infinity after a single dose | 0-840 hours
  Measured in pmol*h/L for insulin 287 following administration of a fixed ratio of NNC0148-0287sema and insulin 287.
Cmax, I287, maximum observed serum insulin 287 concentration after a single dose | 0-840 hours
  Measured in pmol/L for insulin 287 following administration of a fixed ratio of NNC0148-0287sema and insulin 287.
tmax, I287, time to maximum observed serum insulin 287 concentration after a single dose | 0-840 hours
  Measured in hour (h) for insulin 287 following administration of a fixed ratio of NNC0148-0287sema and insulin 287.
AUCSema,0-∞, area under the plasma semaglutide concentration-time curve from 0 hours to infinity after a single dose | 0-840 hours
  Measured in pmol*h/L for semaglutide following administration of a fixed ratio of NNC0148-0287sema and semaglutide.
Cmax,Sema, maximum observed plasma semaglutide concentration after a single dose | 0-840 hours
  Measured in pmol/L for semaglutide following administration of a fixed ratio of NNC0148-0287sema and semaglutide.
tmax,Sema, time to maximum observed plasma semaglutide concentration after a single dose | 0-840 hours
  Measured in hour (h) for semaglutide following administration of a fixed ratio of NNC0148-0287sema and semaglutide.
Number of treatment emergent adverse events | Day 1 (beginning of each period) to day 36 (end of each period)
  Count of events.
Number of hypoglycaemic episodes | Day 1 (beginning of each period) to day 36 (end of each period)
  Count of episodes.
Antibodies for insulin 287: Change in anti-insulin 287 binding antibody levels | Day -1 (pre-dose), Day 36 (end of period)
  Measured as percentage B/T following administration of NNC0148 -0287sema and insulin 287.
Antibodies for insulin 287: Occurrence of anti-insulin 287 binding antibodies | Day 36 (end of period)
  Percentage of events (yes/no) following administration of NNC0148 -0287sema and insulin 287.
Antibodies for insulin 287: Occurrence of anti-insulin 287 binding antibodies cross reacting to human insulin | Day 36 (end of period)
  Percentage of events (yes/no) following administration of NNC0148 -0287sema and insulin 287.
Antibodies for semaglutide: Change in anti-semaglutide binding antibody levels | Day -1 (pre-dose), Day 36 (end of period)
  Measured as percentage B/T following administration of NNC0148 -0287sema
Antibodies for semaglutide: Occurrence of anti-semaglutide binding antibodies | Day 36 (end of period)
  Percentage of events (yes/no) following administration of NNC0148 -0287sema.
Antibodies for semaglutide: Occurrence of anti-semaglutide binding antibodies cross reacting to endogenous glucagon-like peptide-1 (GLP-1) | Day 36 (end of period)
  Percentage of events (yes/no) following administration of NNC0148 -0287sema.
Binding antibodies and in vitro neutralising antibodies (semaglutide only): Anti-semaglutide binding antibody levels | Day 151 (follow-up/end-of-trial visit)
  Measured as percentage B/T.
Binding antibodies and in vitro neutralising antibodies (semaglutide only): Occurrence of anti-semaglutide binding antibodies cross reacting to endogenous GLP-1 | Day 151 (follow-up/end-of-trial visit)
  Percentage of events (yes/no).
Binding antibodies and in vitro neutralising antibodies (semaglutide only): Anti-insulin 287 binding antibody levels | Day 151 (follow-up/end-of-trial visit)
  Measured as percentage B/T.
Binding antibodies and in vitro neutralising antibodies (semaglutide only): Occurrence of anti-insulin 287 binding antibodies cross reacting to human insulin | Day 151 (follow-up/end-of-trial visit)
  Percentage of events (yes/no).
Binding antibodies and in vitro neutralising antibodies (semaglutide only): Occurrence of anti-semaglutide neutralising antibodies | Day 151 (follow-up/end-of-trial visit)
  Percentage of events (yes/no).
Binding antibodies and in vitro neutralising antibodies (semaglutide only): Occurrence of anti-semaglutide neutralising antibodies cross reacting with endogenous GLP-1 | Day 151 (follow-up/end-of-trial visit)
  Percentage of events (yes/no).

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Reporting Anchor and Disclosure (1452), Study Director — Novo Nordisk A/S
Locations (1):
- Profil Institut für Stoffwechselforschung GmbH, Neuss, Germany

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: https://www.novonordisk-trials.com

REFERENCES:
- [Result] Westergaard L, Alifrangis L, Buckley ST, Coester HV, Klitgaard T, Kristensen NR, Nishimura E, Norgreen L, Rocha TMP, Steensgaard DB, Vegge A, Plum-Morschel L. Pharmacokinetic Properties of a Once-Weekly Fixed-Ratio Combination of Insulin Icodec and Semaglutide Compared with Separate Administration of Each Component in Individuals with Type 2 Diabetes Mellitus. Clin Drug Investig. 2024 Nov;44(11):849-861. doi: 10.1007/s40261-024-01405-8. Epub 2024 Nov 3. PMID 39488821